CLINICAL TRIAL: NCT06496399
Title: Psychoeducation Program Given to the Elderly Living Alone at Home in Terms of Some Parameters
Brief Title: Evaluation of the Psychoeducation Program Given to the Elderly Living Alone at Home in Terms of Some Parameters
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kastamonu University (Other)
Responsible Party: Principal Investigator, Zeynep Arabacı, Dr., Kastamonu University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Kastamonu Universitesi
Record Dates: First submitted 2024-04-29; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Nursing Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- trial (Experimental): psychoeducation
  Interventions: Behavioral: psychoeducation
- control (No Intervention): standart care

INTERVENTIONS:
Behavioral: psychoeducation — -The elderly's preferences for art therapy (art activities such as wood painting, creating shapes with mud) will be taken into account.
  2-Expression of emotions through motivational interviewing 3-Conscious Awareness therapy, staying in the moment here and now 4- Hobbies (growing flowers, gardening, handicraft knitting, puzzle solving, card games, chess game, etc., organizing trips, cinema, movie events and so on)
  Arms: trial

SUMMARY:
It was aimed to evaluate the effectiveness of the psychoeducation program given to the elderly living alone at home. In this context, the psychoeducation given was planned to evaluate the effect of the psychological well-being, self-integration and coping levels of the elderly.

DETAILED DESCRIPTION:
The aging process can cause decreases in psychological well-being levels and bring about some mental health problems. It is stated that the most common mental health problems in the elderly are depression, delirium, dementia, anxiety disorders, sleep problems and fear of death. However, factors that negatively affect psychological well-being, such as loneliness experienced in old age and hopeless looking at the future, negatively affect cognitive functions. It can be said that it may affect However, it can be said that the environmental arrangements that can improve the coping channels of elderly individuals and activate them against the changes in old age are very limited.In their studies examining the effect of coping with stress on life satisfaction in the elderly, using optimistic and social support seeking methods while coping with stress increases their life satisfaction. The same study will support intervention programs aimed at increasing the life satisfaction of the elderly. In studies conducted in Turkey, coping skills; Self-confident approach, helpless approach, submissive approach, optimistic approach, seeking social support were determined as self-confident approach, optimistic approach and social support seeking sub-dimensions were determined as effective coping methods, and helpless and submissive approach were determined as ineffective coping methods. It is thought that environmental arrangements that will make elderly individuals happy and prevent them from being alone may be effective in helping them spend more quality time. In this context, psychoeducation will be provided to the elderly living alone at home through regular home visits in order to increase psychological well-being. Within the scope of psychoeducation, the following activities will be planned according to the interests of elderly individuals. 1-Art therapy (the elderly's preferences for artistic pursuits such as wood painting, creating shapes with mud will be taken into account. 2-Expression of emotions through motivational interviewing 3-Conscious Awareness therapy, staying in the present moment 4- Hobbies (growing flowers, gardening, handicraft knitting art, puzzle solving, card games, chess game, etc., organizing trips, cinema, movie events, etc.) With the psychoeducation to be planned, a self-integrative approach will be provided for the elderly person to be happy in the present by accepting the negativities he/she perceives about his/her past, which affects the psychological well-being of the elderly living alone at home. One of the variables is the lack of social support of the elderly. Ensuring the elderly's participation in activities related to their areas of interest by reducing loneliness through home visits will increase both the elderly's coping power and psychological well-being. In the study where they evaluated the psychoeducation given as; They applied psychoeducation consisting of 8 sessions to 42 elderly individuals. Life satisfaction scale after psychoeducation, total score and subscale of healthy lifestyle behaviors scale

It was determined that the mean scores of (nutrition, health responsibility, self-actualization, stress management, interpersonal support and exercise) increased at a statistically significant level.

ELIGIBILITY:
Inclusion Criteria:elderly -

Exclusion Criteria:Those who do not want to participate in the study

-

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2024-12-29 (Estimated); Study Completion 2025-06-29 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Psychoeducation Program in Terms of Some Parameters | 8 week
  psychological well-being, self-integration and coping levels of the elderly

CONTACTS AND LOCATIONS:
Locations (1):
- Zeynep ARABACI, Kastamonu, Turkey (Türkiye)